CLINICAL TRIAL: NCT04547985
Title: Naltrexone Treatment for Prolonged Grief Disorder: A Pilot Study
Brief Title: Naltrexone Treatment for Prolonged Grief Disorder (PGD)
Acronym: PGD
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: We are terminating the study due to low accrual.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20-04021873
Record Dates: First submitted 2020-08-31; First posted 2020-09-14 (Actual); Results first posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Prolonged Grief Disorder
Keywords: Naltrexone
MeSH Terms: conditions — Prolonged Grief Disorder | interventions — Naltrexone; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): 24 randomized patients will take placebo daily for 8 weeks.
  Interventions: Drug: Placebo
- Naltrexone (Active Comparator): 24 randomized patients will take naltrexone daily for 8 weeks
  Interventions: Drug: Naltrexone HCl 50 MG Oral Tablet

INTERVENTIONS:
Drug: Naltrexone HCl 50 MG Oral Tablet — Generic, oral tablet.
  Arms: Naltrexone
Drug: Placebo — Composed of filler material and encapsulated to appear identical to naltrexone.
  Arms: Placebo

SUMMARY:
This is a study to see how effective oral naltrexone is as treatment for prolonged grief disorder (PGD). Participants will take their assigned medication for 8 weeks, with monthly visits to assess symptom severity, social connectedness, and adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older.
2. Lives within a reasonable distance from NYPH for convenient clinic visits.
3. Can speak, read, and write English proficiently.
4. Meet diagnostic criteria for PGD based on the DSM guidelines
5. If a female patient, must agree to use a method of contraception and be willing and able to continue contraception during the first 8 weeks of the study while she is taking the study drug. Female patients who are planning to use oral hormonal contraception during this time must have initiated it at least 2 months prior to the baseline visit.
6. If a male patient, must agree to use a method of contraception and be willing and able to continue contraception during the first 8 weeks of the study while he is taking the study drug.

Exclusion Criteria:

1. Having recently started taking/prescribed medications for any psychiatric illness (e.g. SSRIs for MDD) within the past 3 months; participants who have been taking this medication for longer than 3 months can be included.
2. Having recently started psychotherapy for any psychiatric illness within the past 3 months; participants who have been receiving psychotherapy for longer than 3 months can be included.
3. Prior history of recently active (e.g. within the past 3 months) opioid dependence.
4. Current prescription, non-prescription, or illicit opioid use, (i.e., acute use within the past 14 days or chronic use within the last 30 days), including opioid antagonists for alcohol or opioid dependence, all opioid analgesics, certain cough and cold remedies (e.g., codeine), and certain anti-diarrheal preparations (e.g., loperamide).
5. Possible future use of opioids during the study (e.g. for surgery).
6. Current use of leflunomide (Arava), droperidol (Droleptan), diazepam (Valium), thioridazine (Mellaril, Novoridazine, Thioril), or any other clinically relevant medication that has potential to cause liver injury with concurrent use of naltrexone.
7. Currently pregnant, lactating, or planning to become pregnant during the study.
8. Active hepatitis or liver disease.
9. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels more than one standard deviation (SD) above the upper limit of normal on initial laboratory examination.
10. Screen positive for active suicidal thoughts or behaviors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holly G Prigerson, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kakarala SE, Roberts KE, Rogers M, Coats T, Falzarano F, Gang J, Chilov M, Avery J, Maciejewski PK, Lichtenthal WG, Prigerson HG. The neurobiological reward system in Prolonged Grief Disorder (PGD): A systematic review. Psychiatry Res Neuroimaging. 2020 Sep 30;303:111135. doi: 10.1016/j.pscychresns.2020.111135. Epub 2020 Jul 3. PMID 32629197
- [Derived] Gang J, Kocsis J, Avery J, Maciejewski PK, Prigerson HG. Naltrexone treatment for prolonged grief disorder: study protocol for a randomized, triple-blinded, placebo-controlled trial. Trials. 2021 Feb 1;22(1):110. doi: 10.1186/s13063-021-05044-8. PMID 33522931

RESULTS

PARTICIPANT FLOW:
Period: 1st Clinic Visit (1 Week)
Arm/Group | Placebo | Naltrexone
Started | 6 | 3
Completed | 6 | 3
Not Completed | 0 | 0
Period: 2nd Clinic Visit (4 Weeks)
Arm/Group | Placebo | Naltrexone
Started | 4 | 1
Completed | 4 | 1
Not Completed | 0 | 0
Period: 3rd Clinic Visit (8 Weeks)
Arm/Group | Placebo | Naltrexone
Started | 4 | 1
Completed | 4 | 1
Not Completed | 0 | 0
Period: Follow Up (12 Weeks)
Arm/Group | Placebo | Naltrexone
Started | 4 | 1
Completed | 4 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Naltrexone | Total
Number analyzed (Participants) | 6 | 3 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 1 | 5
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 2 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Prolonged Grief Disorder Symptom Severity as Assessed by Prolonged Grief-13 (PG-13)
Description: Prolonged Grief Disorder (PGD) is a newly defined syndrome that is a specific reaction to the loss of a loved one. Change in PGD symptom severity will be measured by using Prolonged Grief-13-R (PG-13-R), a self-rated scale consisting of 11 items. The validity and reliability of the scale were tested and validated in previous studies.
  Minimum Score: 11 - reflecting the lowest level of PGD symptom severity (distress) Maximum Score: 55 - reflecting the highest level of PGD symptom severity (distress) Diagnostic Criteria PGD symptom severity of ≥30 is the threshold for "syndromal" level PGD.
  Prolonged Grief (PG-13-R) is a diagnostic tool. If a respondent meets the diagnostic criteria for PGD, this suggests that they should seek more thorough evaluation from a mental health professional. Only an in-person assessment by a mental health professional can determine for certain the clinical significance of the reported symptoms, and provide recommendations or referrals for treatment.
Time Frame: Baseline and 8 Weeks
Population: Four participants had dropped out of the study, and therefore, the required data for analysis was not collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Naltrexone
Number analyzed (Participants) | 4 | 1
score on a scale
  Baseline | 44.75 (7.36) | 39 (NA) — Standard Deviation cannot be calculated with a single data point.
  8 Weeks | 25 (11.11) | 40 (NA) — Standard Deviation cannot be calculated with a single data point.

2. Primary Outcome: Change in Prolonged Grief Disorder Symptom Severity as Assessed by Prolonged Grief-13
Description: as for outcome 1
Time Frame: Baseline and 12 weeks
Population: Four participants had dropped out of the study, and therefore, the required data for analysis was not collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Naltrexone
Number analyzed (Participants) | 4 | 1
score on a scale
  Baseline | 44.75 (7.36) | 39 (NA) — Standard Deviation cannot be calculated with a single data point.
  12 Weeks | 25 (11.11) | 41 (NA) — Standard Deviation cannot be calculated with a single data point.

3. Primary Outcome: Change in Number of Participants With Prolonged Grief Disorder as Assessed by Structured Clinical Interview for PGD (SCIP)
Description: Eligibility for the study and change in symptom severity will be measured by SCIP. This structured clinical interview is adapted to the DSM-5-TR criteria for PGD. Interviewers will be trained to standard which will be a κ > 0.8 agreement between trainee and trainer.
Time Frame: Every 4 weeks for 8 weeks
Population: Four participants had dropped out of the study, and therefore, the required data for analysis was not collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Naltrexone
Number analyzed (Participants) | 4 | 1
Participants
  4 weeks | 3 | 1
  8 weeks | 1 | 1

4. Secondary Outcome: Change in Strength of Subjectively Perceived Closeness of a Social Relationship as Measured by the Inclusion of the Other in the Self (IOS) Scale
Description: The Inclusion of Other in the Self (IOS) Scale is a self-reported pictorial tool used to measure the subjectively perceived closeness of a relationship. Respondents choose a pair of seven circles with different degrees of overlap. 1=no overlap; 2=little overlap; 3=some overlap; 4=equal overlap; 5=strong overlap; 6=very strong overlap; 7=most overlap.
  The tool asks respondents to select one of seven pairs of increasingly overlapping circles that best represent their relationship with another, with more overlap signifying a closer relationship. This scale possesses good reliability, with (α=.93) for the entire sample, (α=.87) for family, (α=.92) for friendship, and (α=.95) for romantic relationships. Test-retest reliability shows similar findings, with (α=.83) for the entire sample, (α=.85) for family, (α=.86) for friendship, and (α=.85) for romantic relationships.
  Minimum Score: 1 - reflecting the least amount of overlap Maximum Score: 7 - reflecting the most amount of overlap
Time Frame: Every 4 weeks for 12 weeks
Population: Four participants had dropped out of the study, and therefore, the required data for analysis was not collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Naltrexone
Number analyzed (Participants) | 4 | 1
score on a scale
  4 weeks | 6 (1.15) | 7 (NA) — Standard Deviation cannot be calculated with a single data point.
  8 weeks | 5.25 (1.71) | 7 (NA) — Standard Deviation cannot be calculated with a single data point.
  12 weeks | 3 (5.75) | 5 (NA) — Standard Deviation cannot be calculated with a single data point.

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Placebo | Naltrexone
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3
Other Adverse Events (participants affected / at risk) | 0/6 | 0/3

LIMITATIONS AND CAVEATS:
Due to low accrual, only descriptive statistics are presented.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-18): https://cdn.clinicaltrials.gov/large-docs/85/NCT04547985/Prot_SAP_000.pdf